CLINICAL TRIAL: NCT03805308
Title: The TESLA Trial: Thrombectomy for Emergent Salvage of Large Anterior Circulation Ischemic Stroke
Acronym: TESLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Health Ohio (Other)
Responsible Party: Principal Investigator, Dr. Osama O. Zaidat, Neuroscience and Stroke Medical Director, Mercy Health Ohio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-49
Record Dates: First submitted 2018-12-03; First posted 2019-01-15 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Ischemic Stroke; Thrombectomy
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Thrombectomy

STUDY DESIGN:
Intervention Model Description: TESLA is a pragmatic, phase III, prospective, randomized, open-label, blinded endpoint, multicenter trial. Patients with moderate-large infarcts will be assigned to either best medical management alone (including intravenous recombinant tissue-type plasminogen activator (IV rtPA)) or intra-arterial treatment (IAT) with mechanical thrombectomy added to best medical management. Mechanical thrombectomy will be performed with FDA-approved thrombectomy devices in accordance with the instructions for use (IFU). Patients will be enrolled at up to 25 centers over an anticipated three-year period, with an additional year for trial closeout.
Who Masked: Outcomes Assessor
Masking Description: The patient and the treating physician will be aware of the treatment assignment. Assessment of outcome on NIHSS and mRS will be performed by a certified rater blinded to the treatment allocation. Each site must designate one or more individual(s) to perform these blinded assessments at 24 (16-36) hours, 6 ± 1 days or discharge (whichever is earlier), 30 days ± 7 days, and 90 days ± 30 days from randomization.
  Neuroimaging core lab evaluation will also be assessed in a blinded manner, except for angiographic revascularization grading which will only be performed for the intra-arterial treatment arm.
  Information on treatment allocation will be stored separately from the main study database. An unblinded independent statistician will combine treatment allocation data with the clinical data in order to report to the DSMB. A second blinded statistician will be part of the steering committee.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medical Management (No Intervention): Patients randomized to the medical therapy arm will receive standard medical therapy based on current AHA guidelines.
- Intra-arterial Therapy (Experimental): For patients randomized to the intra-arterial therapy arm, sites will use local protocols for femoral access, sedation, heparin infusion, monitoring, etc. Mechanical thrombectomy will be performed with FDA-approved thrombectomy devices in accordance with the IFU.
  Interventions: Procedure: Intra-arterial Therapy

INTERVENTIONS:
Procedure: Intra-arterial Therapy — Mechanical Thrombectomy is a treatment for stroke that removes clots that block large blood vessels.
  Other Names: Thrombectomy
  Arms: Intra-arterial Therapy

SUMMARY:
The primary objective of the trial is to establish the effectiveness of IAT (versus medical management) in patients with moderate-large infarcts (NCCT ASPECTS 2-5) at baseline, with adaptive enrichment to better define the upper limit of infarct volume for treatment eligibility. Furthermore, the investigators aim to determine whether certain subgroups of patients with large baseline infarcts will have a greater treatment benefit. Finally, the investigators will assess the agreement of ASPECTS scores between site investigators, the core imaging lab, and automated software.

DETAILED DESCRIPTION:
Prospective, randomized, open-label, blinded endpoint study. Patients presenting with symptoms of AIS who have evidence of a moderate-large infarct volume (Non-contrast CT Alberta Stroke Program Early CT score [NCCT ASPECTS] 2-5 in the anterior circulation will be assigned to either best medical management alone (including IV rtPA) or intra-arterial treatment (IAT) with mechanical thrombectomy added to best medical management. Each treated patient will be followed and assessed for 3 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 85 years of age
2. Presenting with symptoms consistent with an acute ischemic stroke
3. Imaging evidence of an anterior circulation occlusion of the Internal Carotid Artery (ICA) terminus and/or Middle Cerebral Artery Main Stem (MCA M1) segment
4. NIHSS score >6 at the time of randomization
5. Ability to randomize within 24 hours of stroke onset
6. Pre-stroke mRS score 0-1
7. Ability to obtain signed informed consent

Imaging evidence of moderate-large infarct defined as:

1. NCCT ASPECTS 2-5

Exclusion Criteria:

1. Females who are pregnant, or those of child-bearing potential with positive urine or serum beta Human Chorionic Gonadotropin (HCG) test
2. Known severe allergy (more than a rash) to contrast media uncontrolled by medications
3. Refractory hypertension (defined as persistent systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg)
4. CT evidence of the following conditions:

   * Midline shift or herniation
   * Evidence of intracranial hemorrhage
   * Mass effect with effacement of the ventricles
5. Computed Tomography Angiography (CTA) evidence suggestive of difficult endovascular access per the treating interventionalist
6. Presence of cervical ICA occlusion (e.g., related to atherosclerotic disease or dissection)
7. Rapidly improving neurological status prior to randomization to NIHSS <6
8. Bilateral strokes or multiple intracranial occlusions
9. Intracranial tumors
10. Known hemorrhagic diathesis, coagulation factor deficiency, or on anticoagulant therapy with an International Normalized Ratio (INR) of >3.0 or Partial Thromboplastin Time (PTT) >3 times of normal
11. Baseline platelet count <30,000 per microliter (µl)
12. Life expectancy less than 90 days prior to stroke onset
13. Participation in another randomized clinical trial that could confound the evaluation of the study
14. Any other condition (in the opinion of the site investigator) that precludes an endovascular procedure or poses a significant hazard to the patient if an endovascular procedure was performed

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-11-18 (Actual)

PRIMARY OUTCOMES:
Utility-weighted 90-day Modified Rankin Score | 90 days post randomization
  Scale used for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. Scale ranges from 0-6 where 0 represents no symptoms and 6 represents death.
  0 = No symptoms at all.
  1. = No significant disability despite symptoms; able to carry out all usual duties and activities.
  2. = Slight disability; unable to carry out all previous activities but able to look after own affairs without assistance.
  3. = Moderate disability requiring some help, but able to walk without assistance.
  4. = Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance.
  5. = Severe disability; bedridden, incontinent, and requiring constant nursing care and attention.
  6. = Death

CONTACTS AND LOCATIONS:
Overall Officials: Albert J Yoo, MD, PhD, Principal Investigator — Texas Stroke Institute; Osama O Zaidat, MD, MS, Principal Investigator — Mercy Health St. Vincent Medical Center
Locations (43):
- United States (43):
  - Baptist Health Center for Clinical Research, Little Rock, Arkansas
  - PIH Health Good Samaritan Hospital and PIH Health Whittier Hospital, Los Angeles, California
  - Pomona Valley Hospital Medical Center, Pomona, California
  - Sutter Institute for Medical Research, Sacramento, California
  - California Pacific Medical Center & Mills Peninsula Medical Center, San Francisco, California
  - Los Robles Hospital and Medical Center, Thousand Oaks, California
  - Providence Saint John's Health Center, Torrance, California
  - Boca Raton Regional Hospital Inc., Boca Raton, Florida
  - University of Miami, Coral Gables, Florida
  - Tenet Health Systems (Delray Medical Center, St. Mary's Medical Center, Palmetto General Hospital), Delray Beach, Florida
  - Orlando Health Inc., Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Wellstar Health System, Inc., Marietta, Georgia
  - The University of Chicago, Chicago, Illinois
  - Northwestern University, Evanston, Illinois
  - AMITA Resurrection Medical Center and AMITA Saint Joseph Medical Center, Lisle, Illinois
  - Central DuPage Hospital Association d/b/a Northwestern Medicine Central DuPage Hospital, Winfield, Illinois
  - Lutheran Medical Group, Fort Wayne, Indiana
  - Munster Medical Research Foundation, Munster, Indiana
  - The University of Iowa, Iowa City, Iowa
  - Baptist Healthcare System Inc. d/b/a Baptist Health Lexington, Lexington, Kentucky
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - University of Massachusetts, Worcester, Massachusetts
  - McLaren Health Care Corporation, Grand Blanc, Michigan
  - Western Michigan University Homer Stryker MD School of Medicine and Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - SSM Health DePaul Hospital, Bridgeton, Missouri
  - Saint Louis University, St Louis, Missouri
  - The Community Hospital Group Inc. t/a JFK Medical Center, Edison, New Jersey
  - Rutgers The State University, Piscataway, New Jersey
  - University of Buffalo, Buffalo, New York
  - Feinstein Institute for Medical Research, Northwell, Manhasset, New York
  - ProMedica Toledo Hospital, Toledo, Ohio
  - Mercy Health St. Vincent Medical Center, Toledo, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - Texas Tech University of Health Sciences, El Paso, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Texas Stroke Institute, Plano, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Valley Medical Center, Renton, Washington
  - West Virginia University, Morgantown, West Virginia
  - Aurora Research Institute, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No
All shared data will be aggregate.

REFERENCES:
- [Derived] Writing Committee for the TESLA Investigators; Yoo AJ, Zaidat OO, Sheth SA, Rai AT, Ortega-Gutierrez S, Given CA 2nd, Zaidi SF, Grandhi R, Cuellar H, Mokin M, Katz JM, Alshekhlee A, Taqi MA, Ansari SA, Siddiqui AH, Barazangi N, English JD, Maud A, Kirmani J, Gupta R, Yavagal DR, Tarpley J, Pandya DJ, Cress MC, Dharmadhikari S, Asif KS, Kass-Hout T, Puri AS, Janjua N, Majjhoo AQ, Badruddin A, Edgell RC, Khatri R, Morgan L, Razak A, Zha A, Khandelwal P, Mueller-Kronast N, Rivet DJ, Wolfe T, Snelling B, Sultan-Qurraie A, Lin SP, Khangura R, Spiotta AM, Bhuva P, Salazar-Marioni S, Lin E, Tarabishy AR, Samaniego EA, Kolikonda MK, Jumaa MA, Reddy VK, Sharma P, Berkhemer OA, van Doormaal PJ, van Es ACGM, van Zwam WH, Emmer BJ, Beenen LF, Majoie CBLM, Buderer N, Detry MA, Bosse A, Graves TL, Saunders C, Elijovich L, Jadhav A, Patterson M, Slight H, Below K, Al Kasab S; TESLA Investigators. Thrombectomy for Stroke With Large Infarct on Noncontrast CT: The TESLA Randomized Clinical Trial. JAMA. 2024 Sep 23;332(16):1355-66. doi: 10.1001/jama.2024.13933. Online ahead of print. PMID 39374319
- [Derived] Roaldsen MB, Jusufovic M, Berge E, Lindekleiv H. Endovascular thrombectomy and intra-arterial interventions for acute ischaemic stroke. Cochrane Database Syst Rev. 2021 Jun 14;6(6):CD007574. doi: 10.1002/14651858.CD007574.pub3. PMID 34125952